CLINICAL TRIAL: NCT01807143
Title: Observational - Gene Discovery in Osteosarcoma
Brief Title: Genetic Biomarkers in Tissue Samples From Patients With Osteosarcoma
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AOST10B1; NCI-2013-00124 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-03-06; First posted 2013-03-08 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Osteosarcoma
MeSH Terms: conditions — Osteosarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Correlative studies: Tissue samples are analyzed for translocations and deletions and analyzed using PCR or FISH.
  Interventions: Other: laboratory biomarker analysis

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This clinical trial studies genetic biomarkers in tissue samples from patients with osteosarcoma. Studying samples of tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer

DETAILED DESCRIPTION:
Study Subtype: Ancillary/Correlative Observational Study Model: Cohort Time Perspective: Retrospective Biospecimen Retention: Samples With DNA Biospecimen Description: Tissue Study Population Description: Samples from the COG Sampling Method: Non-Probability Sample

PRIMARY OBJECTIVES:

I. To use PET sequencing to analyze DNA from ten human primary osteosarcoma samples, along with matched normal tissue where available.

OUTLINE:

Tissue samples are analyzed for translocations and deletions and analyzed using polymerase chain reaction (PCR) or fluorescence in situ hybridization (FISH).

ELIGIBILITY:
Inclusion Criteria:

* Samples from the COG tissue repository

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Osteosarcoma
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2010-01; Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Mapping and filtering of paired tags | Up to 2 years
  Mapping of paired tags to reference genomes to identify aberrant pairs, caused by translocations, insertions, deletions and inversions.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Gorlick, MD, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Monrovia, California, United States